CLINICAL TRIAL: NCT01962740
Title: Serial Evaluation of Drug-Eluting Stents Using OCT
Brief Title: Serial Evaluation of Drug-Eluting Stents Using OCT (STRUT-OCT)
Acronym: STRUT-OCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible patients
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shuaib Abdullah, MD, Cardiologist; Assistant Professor, Division of Cardiology, Internal Medicine, UT Southwestern Medical School, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-043
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Drug Eluting Stents (DES); Percutaneous Coronary Intervention (PCI); Uncovered and Malapposed Stent Struts; Optical Coherence Tomography (OCT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Xience EES (Active Comparator): This arm of patients will receive Xience Everolimus Eluting Stents(EES) as part of their clinically indicated PCI procedure and they will undergo Optical Coherence Tomography Imaging
  Interventions: Device: Drug-eluting stent implantation
- Resolute Integrity ZES (Active Comparator): This arm of patients will receive Resolute Integrity Zotaralimus Eluting Stents (ZES) as part of their clinically indicated PCI procedure and they will undergo Optical Coherence Tomography Imaging
  Interventions: Device: Drug-eluting stent implantation
- Promus Element EES (Active Comparator): This arm of patients will receive Promus Element Everolimus Eluting Stents (EES) as part of their clinically indicated PCI procedure and they will undergo Optical Coherence Tomography Imaging
  Interventions: Device: Drug-eluting stent implantation

INTERVENTIONS:
Device: Drug-eluting stent implantation

SUMMARY:
The study is proposed as a 48-patient randomized-controlled pilot study that will use Optical Coherence Tomography (OCT) imaging to compare stent strut coverage and malapposition of three second-generation Drug Eluting Stents (DES) [Xience EES (Abbott Vascular, Santa Clara, CA), Resolute Integrity ZES (Medtronic, Minneapolis, MN) and Promus Element EES (Boston Scientific, Natick, MA)] at 6 weeks post implantation.

Study Hypothesis is that the rates of stent strut coverage and malapposition of the Xience EES, Promus EES and will be similar to each other and improved (higher rates of stent strut coverage and lower rates of malapposition) compared to the Resolute ZES at 6 weeks post-implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Clinical need for percutaneous coronary intervention using either a Xience, Promus Element, or Resolute Integrity drug-eluting stent using optical coherence tomography optimization
3. Native coronary artery de novo lesion with ≥70% angiographic percent diameter stenosis by visual estimation
4. Target vessel reference diameter between 2.5 and 4.0 mm by visual estimate
5. Target lesion ≤28 mm in length by visual estimate
6. Agree to participate and provide informed consent

Exclusion Criteria:

1.Presentation with acute ST-elevation myocardial infarction (defined as electrocardiographic (ECG) ST-elevation ≥ 2 mm in 2 or more contiguous ECG leads along with symptoms compatible with ischemia)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Stent Strut Coverage | 6 weeks post-implantation
Stent Strut Malapposition | 6 weeks post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Shuaib Abdullah, MD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No